CLINICAL TRIAL: NCT04065620
Title: Evaluation of Ambulatory Blood Pressure Measurement Related Hemodynamic Biomarkers On the Progression of Heart Failure With Preserved Ejection Fraction
Brief Title: Ambulatory Blood Pressure in HFPEF Outcomes Global Registry
Acronym: HFPEFGlobal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Miguel Camafort, Miguel Camafort-Babkowski MD PhD. Principal Investigator. Consultant Physician, Internal Medicine department. Heart Failure Unit ., Hospital Clinic of Barcelona
Other Study IDs: MDIUB201901
Record Dates: First submitted 2019-07-25; First posted 2019-08-22 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Arterial Hypertension; Frailty Syndrome; Comorbidities and Coexisting Conditions
Keywords: Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Hypertension; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ambulatory blood pressure measurement — 24-hour ABPM will be made using validated devices, following ABPM device should be programmed to take measurements every 30 minutes . Patients will be instructed in their use. Periods of activity and rest will be pre-determined in short windows: for Asian and European Countries daytime period will be defined between 10:00 and 8:00 pm; and night-time period between 00:00 am and 6:00 am. For Latin American Countries daytime period will be defined between 08:00 and 06:00 pm; and night-time period between 00:00 am and 6:00 am. For Africa daytime period will be defined between 08:00 and 06:00 pm; and night-time period between 11 PM and 5 AM In addition, the duration of ABPM (hours), the percentage of valid readings, and the mean SBP/DBP values during periods of activity, rest and in 24 hours will be recorded. Records with a duration <24 hours, those without one good reading per hour and those with <70% of satisfactory readings will be excluded
  Other Names: home blood pressure measurement; Short Physical Performance Battery

SUMMARY:
Heart failure and preserved ejection fraction (HFPEF) is a disease with increasing prevalence world wide. Due to its etiological and prognostic relationship with hypertension, it is highly interesting to know the characteristics and influence of Blood pressure levels and of the hemodynamic biomarkers, measured by Ambulatory Blood Pressure measurement in the outcome of patients with (HF-PEF), defined by the risk of cardiovascular morbidity and mortality (hospital re-admissions, emergency room visits, functional decline and mortality). The investigators consider other factors such as Frailty, comorbidities, and the baseline functional capacity to asses the prognostic value.

DETAILED DESCRIPTION:
The prognosis of patients with heart failure and preserved ejection fraction (HF-PEF), defined by the risk of cardiovascular morbidity and mortality (hospital re-admissions, emergency room visits, functional decline and mortality), depends on multiple factors such as Frailty, comorbidities, BP values, hemodynamic parameters and the baseline functional capacity. Correct definition of these prognostic factors may help define more effective management strategies This is a Prospective observational cohort study, aimed to identify prognostic factors of readmission for heart failure or death in patients with HF-PEF.

Patients with stable HF-PEF will be included monitoring will be by telephone or personal interview every 3 months for at least one year.Specific data on HF will be collected directly from the patient, or from the computerized medical record, with the objective of determining different aspects of HF.

An echocardiogram performed 6 months before inclusion in the case of known HF, or up to 3 months after inclusion, will be considered valid. Parameters collected will include ejection fraction, dimensions of the atrium and ventricle and variables of diastolic dysfunction. ( The procedures for BP measurement, will be according to the ESH/ESC 2018 guidelines, All patients included in the study should have a 12 lead rest EKG performed at study inclusion. Data will be required on renal function (creatinine and glomerular filtration rate and microalbuminuria), lipid parameters (cholesterol: total, HDLc, LDLc,), baseline glucose, glycated hemoglobin (HbA1c), liver biology (GOT, GPT, GGT), albumin and prealbumin, blood cell count, Ferritin and Transferrin saturation rate, natriuretic peptides.

In some centres blood sample will be collected to a further evaluation of biomarkers.

24-hour ABPM will be made using validated devices, ABPM device should be programmed to take measurements every 30 minutes . Patients will be instructed in their use. Periods of activity and rest will be pre-determined in short windows: In addition, the duration of ABPM (hours), the percentage of valid readings, and the mean SBP/DBP values during periods of activity, rest and in 24 hours will be recorded. Records with a duration <24 hours, those without one good reading per hour and those with <70% of satisfactory readings will be excluded. ABPM will be performed at baseline and at the final visit HBPM should be done by a trained individual (the patient or anyone else), with equipment validated, calibrated and provided with memory.

Only validated semiautomatic oscillometric arm cuff devices are recommended for these measurements. The functional status will be determined using the Barthel index, Cognitive impairment will be tested following the Montreal Cognitive Assessment with local adaptations.

The diagnosis of frailty will be made using the Short Physical Performance Battery In a subset of centres a 24H ambulatory ECG recording will be performed using a standard recording unit and automatically analyzed by a PC-based Holter system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous diagnosis of HF-PEF, defined by:
* At least a previous hospitalization due to heart failure
* Left ventricular ejection fraction (LVEF) ≥45% by echo during screening epoch, or within 6 months prior to study entry.
* Symptom(s) of heart failure (HF) and requiring, at least 30 days prior to study entry, hospitalization, or consultation to emergency room .
* Current symptom(s) of HF
* Structural heart disease documented by echocardiogram, namely septal or posterior wall thickness >=1.1 cm) or LA enlargement (i.e., width >=3.8 cm, length >=5.0 cm, area >=20 cm2, volume >=55 ml, or volume index >=29 ml/m
* Elevated NT-proBNP defined as NT-proBNP >200 pg/ml if the patient had been hospitalized for HF within the past 9 months or >300 pg/ml if not so.

Clinical and hemodynamic stability for at least 4 weeks before study inclusion, defined as stable treatment or functional class for at least 4 weeks before study inclusion, (changes in diuretic dosification are not considered as unstable treatment).

Exclusion Criteria:

* Any prior measurement of LVEF ≤ 40%.
* Acute coronary syndrome (including MI), cardiac surgery, other major CV surgery within 3 months , urgent percutaneous coronary intervention or limb amputation due to peripheral arterial disease or Stroke within 3 months or and elective PCI within 30 days prior to entry.
* Current acute decompensated HF requiring therapy.
* Changes in antihypertensive treatment (class type or dose) 4 weeks before inclusion, excluding changes in diuretics due to congestion.
* Alternative reason for shortness of breath such as: significant pulmonary disease or severe COPD, haemoglobin (Hgb) <10 g/dl, or body mass index (BMI) > 40 kg/m2.
* Systolic blood pressure (SBP) ≥ 180 mmHg or DBP ≥ 110 mmHg at entry.
* Patients with severe chronic renal disease, defined as GFR <15 ml/min or haemodialysis.
* Inability to understand the study and participate voluntarily
* Patients diagnosed with cancer in the previous 12 months, and requiring treatment, at the time of study inclusion.
* Patients diagnosed with systemic autoimmune disease (lupus, vasculitis . . .)
* Patients not able to perform an ambulatory blood pressure measurement namely working at night, or patients with tachyarrhythmia.

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stable HF-PEF
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Morbimortality | 1 year
  Influence of ambulatory Blood pressure measurement derived biomarkers on the incidence of the composite of the number of hospital readmission due to HF, number of CV and non CV death or number of patients with functional decline in patients with HF-PEF

SECONDARY OUTCOMES:
Readmission | 1 year
  Influence of hemodynamic biomarkers of BP measured by ABPM on the number of new hospital readmissions in patients with HF-PEF.
CV mortality | 1 year
  Influence of hemodynamic biomarkers of Blood pressure measured by ABPM on the number of patients with HFPEF presenting CV and non CV death.
Functional decline | 1 year
  Influence of hemodynamic biomarkers of Blood pressure measured by ABPM on the functional decline in patients with HF-PEF, measured by changes in the Barthel index scale
Cognitive decline | 1 year
  Influence of hemodynamic biomarkers of Blood pressure measured by ABPM on the functional decline in patients with HF-PEF, measured by changes in the Montreal Cognitive assessment scales
Frailty | 1 year
  Influence of hemodynamic biomarkers of Blood pressure measured by ABPM on the functional decline in patients with HF-PEF, measured by changes in the short performance battery scale

OTHER OUTCOMES:
Influence of cognitive impairment on outcomes in HFPEF | 1 year
  incidence of the composite of the number of hospital readmission due to HF, number of CV and non CV death or number of patients with functional decline in patients with HF-PEF related to baseline Montreal Cognitive Assessment scale Values
Influence of frailty on outcomes in HFPEF | 1 year
  incidence of the composite of the number of hospital readmission due to HF, number of CV and non CV death or number of patients with functional decline in patients with HF-PEF related to baseline Short Physical Performance Battery Values

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Camafort-Babkowski, MD PhD, Study Director — Internal Medicine Department. Hospital Clinic. University of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided